CLINICAL TRIAL: NCT03693560
Title: The Effect of Adding Vildagliptin Versus Glimepiride to Metformin on Markers of Inflammation, Thrombosis, and Atherosclerosis in Diabetic Patients With Symptomatic Coronary Artery Diseases
Brief Title: Effect of Adding Vildagliptin vs Glimepiride to Metformin on Inflammation's Markers in Type-2 Diabetic Patients With CAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Principal Investigator, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: vildaglipitin in CAD
Record Dates: First submitted 2018-09-25; First posted 2018-10-03 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Tablets; Metformin; glimepiride

STUDY DESIGN:
Intervention Model Description: All enrolled patients will be mentioned as two groups; Group I (n=40) are patients who the endocrinologist prescribed them vildagliptin plus their metformin to control their blood sugar level. Group II (n=40) are patients who the endocrinologist prescribed them glimepiride plus their metformin.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vildagliptin / metformin (Experimental): Group I (n=40) are patients who are taking vildagliptin 50 mg oral tablet plus their metformin1000 mg oral tablet to control their blood sugar level.
  Interventions: Drug: Vildagliptin 50 mg Oral Tablet; Drug: Metformin 1000 mg Oral Tablet
- glimepiride / metformin. (Experimental): Group II (n=40) are patients who are taking Glimepiride 4 mg oral tablet plus their metformin1000 mg oral tablet to control their blood sugar level.
  Interventions: Drug: Metformin 1000 mg Oral Tablet; Drug: Glimepiride upto 4 mg Oral Tablet

INTERVENTIONS:
Drug: Vildagliptin 50 mg Oral Tablet — Patients who the endocrinologist prescribed them Vildagliptin 50 mg Oral Tablet plus their Metformin 1000 mg Oral Tablet to control their blood sugar level.
  Other Names: Galvus 50 mg
  Arms: vildagliptin / metformin
Drug: Metformin 1000 mg Oral Tablet — Patients with Coronary artery diseases.and uncontrolled Diabetes Mellitus type 2 who's taking Metformin 1000 mg Oral Tablet only will be enrolled from endocrinology clinic.
  Other Names: Glucophage 1000 mg
Drug: Glimepiride upto 4 mg Oral Tablet — Patients who the endocrinologist prescribed them Glimepiride 4 mg oral tablet plus their Metformin 1000 mg Oral Tablet
  Other Names: Amaryl 4 mg
  Arms: glimepiride / metformin.

SUMMARY:
The aim of this study is to evaluate the effect of adding Vildagliptin versus Glimepiride to Metformin on markers of inflammation, thrombosis, and atherosclerosis in diabetic patients with symptomatic Coronary artery diseases.

The pre-specified established biological markers of inflammation, thrombosis, and atherosclerosis will include: Interleukin 1 beta (IL-1 beta)), hs-CRP, Atherogenic index and coronary risk index, Lipid profile. and adiponectin levels..

DETAILED DESCRIPTION:
The study is designed as a single-center, randomized, double-blinded, clinical trial to provide evidence on the effects of vildagliptin on key biomarkers of atherothrombosis and inflammation. The investigators plan to prospectively enroll 80 patients with proven coronary artery disease ,Diabetes type2 and randomize them in a 1:1 ratio to either vildagliptin-metformin therapy (n=40) or glimepiride /metformin therapy (n=40).

1. All participants agreed to take part in this clinical study and provide informed consent.
2. Patients with Coronary artery diseases.and uncontrolled Diabetes type2 who's taking metformin only will be enrolled (n=80) from endocrinology clinic at Alexandria Armed Forces hospital.
3. Complete physical, laboratory, radiological assessment will be done for all patients to exclude any signs of inflammation or thrombosis.
4. Serum samples will be collected for measuring the biomarkers.
5. All enrolled patients will be mentioned as two groups; Group I (n=40) are patients who the endocrinologist prescribed them vildagliptin plus their metformin to control their blood sugar level. Group II (n=40) are patients who the endocrinologist prescribed them glimepiride plus their metformin.
6. All patients will be followed up during 3 months' period.
7. At the end of 3 months on the new regimen, steps 4 and 5 will be repeated.
8. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
9. Measuring outcome: The primary outcome is the change of serum levels of the measured inflammatory markers after 3 months.
10. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Type II-diabetes mellitus on metformin who are planned to be managed with vildagliptin or glimepiride plus metformin at the time of inclusion.
* Symptomatic Coronary Artery Diseases. (>30 days).

Exclusion Criteria:

* Hepatic impairment.
* Active malignancy.
* Planned surgical intervention.
* Any signs of hypersensitivity or contraindication to study drugs developed.
* Any patient with any signs of active infection or thrombosis at the time of assessment.
* Addition of any antidiabetic medications or insulin during follows up.
* Chronic inflammatory disease (i.e. inflammatory bowel disease, lupus, inflammatory arthritis, rheumatoid arthritis) or chronic infection (i.e. chronic diabetic foot infection).
* Clinically advanced congestive heart failure - New York Heart Association III-IV
* Severe left ventricular dysfunction (LVEF<30%) with New York Heart Association II or any New York Heart Association class with documented recent heart failure decompensation (<3 months)
* Severe stable cardiac angina Community Competence Scale III - IV or Unstable angina
* Pregnancy, lactation or child-bearing potential.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Change in markers of athero-thrombosis and inflammation ( interleukin (IL)-1 beta). | Baseline and 3 months
  A-Change in interleukin (IL)-1 beta (IL-1ß) level will be determined by Enzyme-linked immunosorbent assay (ELISA). (unit: Picogram/milliliter pg/ml).
Change in High sensitivity C-reactive protein (hsCRP) level. | Baseline and 3 months
  A- High sensitivity C-reactive protein (hsCRP) level will be determined by nephelometric procedure.(unit: mg/L)
Change in Adiponectin level. | Baseline and 3 months
  A- Adiponectin level will be determined by Enzyme-linked immunosorbent assay (ELISA)..(unit: mg/L)

SECONDARY OUTCOMES:
Change in Lipid profile | Baseline and 3 months
  A-Change inTriglycerides (TGs). (Unit : milligrams per deciliter (mg/dL)) B-Change in total cholesterol (TCH). (Unit : milligrams per deciliter (mg/dL)) C-Change in high-density lipoprotein (HDL-C). (Unit : milligrams per deciliter (mg/dL)) D-change in Low density lipoprotein cholesterol (LDL-C). (Unit : milligrams per deciliter (mg/dL))
Percent Change in ( Low-density lipoprotein (LDL) cholesterol / High-density lipoprotein (HDL) cholesterol ) for each patient before and after 3 months combination treatment for each group . | Baseline and 3 months
  Percent Change in (Low-density lipoprotein (LDL) cholesterol/High-density lipoprotein (HDL) cholesterol) =(combination treatment value - baseline value) / baseline value*100
Change in Hemoglobin A1c (HbA1c). | Baseline and 3 months
  A-Change in Hemoglobin A1c (HbA1c) by ion exchange method.(Unit : percent )
Percent Change in (total cholesterol / High-density lipoprotein (HDL) cholesterol) for each patient before and after 3 months combination treatment for each group . | Baseline and 3 months
  Percent Change in (total cholesterol / High-density lipoprotein (HDL) cholesterol) =(combination treatment value - baseline value) / baseline value*100

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Omran, PhD, Study Director — Faculty of Pharmacy - Damanhour University.; Tarek Mostafa, PhD, Study Director — Tanta University; Ahmed skokry, PhD, Study Director — Alex.Armed Forces Hospital.; Rehab Werida, PhD, Study Director — Faculty of Pharmacy - Damanhour University.; Mahmoud kabel, Principal Investigator — Faculty of Pharmacy - Damanhour University
Locations (1):
- Faculty of Pharmacy - Damanhour University., Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klempfner R, Leor J, Tenenbaum A, Fisman EZ, Goldenberg I. Effects of a vildagliptin/metformin combination on markers of atherosclerosis, thrombosis, and inflammation in diabetic patients with coronary artery disease. Cardiovasc Diabetol. 2012 Jun 6;11:60. doi: 10.1186/1475-2840-11-60. PMID 22672501
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] Yin M, Sillje HH, Meissner M, van Gilst WH, de Boer RA. Early and late effects of the DPP-4 inhibitor vildagliptin in a rat model of post-myocardial infarction heart failure. Cardiovasc Diabetol. 2011 Sep 28;10:85. doi: 10.1186/1475-2840-10-85. PMID 21955567
- [Background] Younis A, Eskenazi D, Goldkorn R, Leor J, Naftali-Shani N, Fisman EZ, Tenenbaum A, Goldenberg I, Klempfner R. The addition of vildagliptin to metformin prevents the elevation of interleukin 1ss in patients with type 2 diabetes and coronary artery disease: a prospective, randomized, open-label study. Cardiovasc Diabetol. 2017 May 22;16(1):69. doi: 10.1186/s12933-017-0551-5. PMID 28532406
- [Background] Derosa G, Maffioli P, Ferrari I, Mereu R, Ragonesi PD, Querci F, Franzetti IG, Gadaleta G, Ciccarelli L, Piccinni MN, D'Angelo A, Salvadeo SA. Effects of one year treatment of vildagliptin added to pioglitazone or glimepiride in poorly controlled type 2 diabetic patients. Horm Metab Res. 2010 Aug;42(9):663-9. doi: 10.1055/s-0030-1255036. Epub 2010 Jun 17. PMID 20560108
- [Background] Kazemi T, Hajihosseini M, Moossavi M, Hemmati M, Ziaee M. Cardiovascular Risk Factors and Atherogenic Indices in an Iranian Population: Birjand East of Iran. Clin Med Insights Cardiol. 2018 Feb 20;12:1179546818759286. doi: 10.1177/1179546818759286. eCollection 2018. PMID 29497341
- [Background] El-Mesallamy HO, Hamdy NM, Salman TM, Mahmoud S. Adiponectin and E-selectin concentrations in relation to inflammation in obese type 2 diabetic patients with coronary heart disease(s). Minerva Endocrinol. 2011 Sep;36(3):163-70. PMID 22019747
- [Result] Werida R, Kabel M, Omran G, Shokry A, Mostafa T. Comparative clinical study evaluating the effect of adding Vildagliptin versus Glimepiride to ongoing Metformin therapy on diabetic patients with symptomatic coronary artery disease. Diabetes Res Clin Pract. 2020 Dec;170:108473. doi: 10.1016/j.diabres.2020.108473. Epub 2020 Sep 28. PMID 33002553

DOCUMENTS (1):
  • Study Protocol (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03693560/Prot_000.pdf